CLINICAL TRIAL: NCT02426424
Title: Effect Of Early C-PAP Treatment For Sleep Apnea On Rehabilitation Of Stroke Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to have funding to perform the trial
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Gal Ifergane MD, Head of Neurology Department, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR-0305-14-ctil
Record Dates: First submitted 2014-12-24; First posted 2015-04-27 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Sleep Apnea; Stroke
Keywords: c-PAP
MeSH Terms: conditions — Sleep Apnea Syndromes; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigatory 1 (Experimental): The sleep study will be performed via Watchpat during the index hospitalization with acute stroke. Following the diagnosis of sleep apnea, patients will be treated with C-PAP both during the hospital stay and after discharge for three months.
  Interventions: Device: Watchpat; Device: CPAP
- Investigatory 2 (Experimental): The sleep study will be performed via Watchpat at home three months after hospitalization with acute stroke. Following the diagnosis of sleep apnea, patients will be treated with C-PAP for three months.
  Interventions: Device: Watchpat; Device: CPAP

INTERVENTIONS:
Device: Watchpat — WatchPAT ™ is an FDA-approved portable diagnostic device that uses the most innovative technology to ensure the accurate screening, detection, and the follow-up treatment of sleep apnea.
Device: CPAP — Continuous positive airway pressure (CPAP) is a form of positive airway pressure ventilator, which applies mild air pressure on a continuous basis to keep the airways continuously open in a patient who is able to breathe spontaneously on his or her own.

SUMMARY:
This is a prospective randomized open label trial with control-to-treatment cross-over. The investigators wish to assess the effectiveness and safety of immediate detection and treatment for Sleep Apnea in Stroke patients. The investigators hypothesize that in patients with acute ischemic stroke a sleep apnea treatment by CPAP will result in a better neurological outcome and more successful rehabilitation.

The study will enroll 140 subjects which will be randomized into one of two arms:

* Investigational - The sleep study will be performed during the index hospitalization with acute stroke. Following the diagnosis of sleep apnea, patients will be treated with C-PAP both during the hospital stay and after discharge.
* Control group -Will receive standard medical care. Patients will undergo sleep study at 3 months following discharge and patients diagnosed with sleep apnea will be treated with C-PAP.

DETAILED DESCRIPTION:
Patients eligible to be enrolled in this study are patients admitted to the Department of Neurology due to acute ischemic stroke up to 72 hours from the start of the stroke symptoms.

After receiving written informed consent from the patient, patients will be randomized into the intervention and control groups (1:1). The intervention group will be tested for sleep apnea and C-PAP treatment will be initiated during the initial hospitalization. The control group will receive standard medical care. Control group patients will undergo sleep study at 3 months following discharge and patients diagnosed with sleep apnea will be treated with C-PAP.

All subjects:

* At the baseline, physical examination MRS and NIHSS will be performed by the neurologist.
* Sleep testing at the baseline with mobile sleep lab device (Watch PAT)
* Four questionnaires will be administered for all patients: Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), quality of life (SF36), depression scale (Beck).
* Blood sample will be taken for CRP, TNF-alpha, IL-6 and IL1 beta, VEGF, HBA1C, LDL and markers of endothelial dysfunction. These blood tests will be repeated at 3 and 6 months.
* At discharge from the Neurology Department, 3 months and 6 months all patients will undergo NIHSS assessment.
* Patients will be referred to the Soroka stroke clinic with rehabilitation program.
* All patients will undergo 3 brain MRI scans, at baseline hospitalization, 3 and 6 months after.

Intervention group:

* In the intervention group, the mobile sleep lab device (Watch PAT) will be used to identify patients with sleep apnea.
* Treatment phase: Patients with (apnea hypopnea index) AHI≥15 will receive an in-hospital treatment with CPAP and continue CPAP treatment following discharge. The CPAP parameters will be titrated during the hospital stay.

Control group:

* Patients will receive standard medical care. At three months, patients will undergo home sleep test with Watch-PAT device.
* Patients with (apnea hypopnea index) AHI≥15 will receive CPAP treatment with titration at home.

TRIAL PROCEDURES 1. Patients eligible to be enrolled in this study are patients admitted to the Neurology Department due to stroke up to 72 hours after the showing of stroke symptoms.

2. At the baseline, physical examination, MRS and NIHSS will be performed by one of the Neurology Department doctors.

3. After receiving written informed consent from the patient, patients will be divided into 2 groups. Study group will have detection and treatment in 72 hours after stroke. Control group will have detection and treatment 3 months after stroke.

STUDY AND CONTROL GROUP

1. The patient will answer four questionnaires: Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), "quality of life" (SF36) and "depression scale" (beck).
2. Next, the mobile sleep lab device (Watch PAT) will be placed on the patient's finger which will provide the apnea-hypopnea Index (AHI) and respiratory disturbance index (RDI).
3. Blood samples for circulating inflammatory biomarkers and endothelial dysfunction will be performed in the morning. Four tubes of peripheral venous blood will be drawn. Every study patient will be tested for the presence of pro-inflammatory state. Specifically, the investigators will measure the presence of high sensitive C Reactive Protein (CRP) and centrifuged sera will be tested (by ultra- sensitive ELISA), for levels of circulating TNF-alpha, IL-6 and IL1 beta. Sera will also be tested for vascular endothelial growth factor (VEGF) and markers of endothelial dysfunction; P-selectin. LDL, HBA1C.
4. At discharge from the Neurology Department, the patient will undergo NIHSS assessment.
5. Half of patients randomly chosen will be asked to join an "early treatment" group for 6 months of C-PAP treatment. Patients from the other half will be asked for C-PAP treatment at 3 months (late intervention).
6. All four questionnaires will be completed by all patients at the end of the follow up period.
7. MRI scan will be done at three points: CVA admission, 3 and 6 months after.
8. Six months after baseline hospitalization, patients from both groups will answer four questionnaires: Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), "quality of life" (SF36) and "depression scale" (beck).

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18.
2. Admitted to the Neurology Department due to acute ischemic stroke.
3. Able to sign informed consent.
4. Admission NIHSS 6-12.

Exclusion Criteria:

1. Stroke symptom onset more than 72 hours prior to the enrollment
2. Transient Ischemic Attack.
3. Chronic pulmonary disease requiring home oxygen treatment.
4. History of C-PAP treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
NIHSS change from the baseline to 3 months | 3 months
  Change in the NIHSS score from admission to three months

SECONDARY OUTCOMES:
NIHSS change score from admission to discharge from the Neurology Department. | 3 months
NIHSS score change from admission to 6 months following hospitalization | 6 months
NIHSS score change from three to six months following hospitalization | 6 month
Prevent recurrent strokes at 6 months | 6 months
Analyse the composite of cardiovascular events at 6 months (acute myocardial infarction, coronary revascularization, death or recurrent stroke) | 6 months
Evaluate new MRI ischemic lesions between 3 MRI scans. | 6 months
Change Epworth Sleepiness Scale (ESS) at 3 and 6 months from the baseline | 6 months
Change quality of life (SF36) at 3 and 6 months from the baseline | 6 months
Change depression scale (Beck) at 3 and 6 months from the baseline | 6 months
Change number of severe adverse events (SAE) at 3 months | 3 months